CLINICAL TRIAL: NCT05368337
Title: Feasibility and Usability of Intrinsic Capacity Monitoring With Eforto and Its Predictive Value for Health Outcomes in Older Community-dwelling Persons
Acronym: FORTO 2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); INNOVIRIS (Unknown); AAL (Unknown)
Responsible Party: Principal Investigator, Prof. Ivan Bautmans, Professor, Vrije Universiteit Brussel
Other Study IDs: FORTO 2.0
Record Dates: First submitted 2022-02-22; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Frailty
Keywords: muscle fatigability; self-monitoring; prevention; self-perceived fatigue
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this study, 160 community-dwelling older adults (65 years and older) will be provided with an eforto® system to self-monitor their muscle fatigability and self-perceived fatigue for 2 consecutive days per week during 12 months (if needed with assistance by an informal caregiver). Preferably, the participants will use their own smartphone because mitigating smartphone-use-related issues.

The aims of the study are:

1. to evaluate the usability and feasibility of self-monitoring intrinsic capacity by using the eforto® system in the home setting.
2. to investigate if changes and variability in intrinsic capacity as measured with eforto® (muscle fatigability and self-perceived fatigue), are related to changes in frailty status, functional independency and quality of life.
3. to explore whether intrinsic capacity as measured with eforto® (muscle fatigability and self-perceived fatigue) is related to circulating inflammatory biomarkers.

DETAILED DESCRIPTION:
Investigational device:

The eforto® system was developed based on approximatively 20 years of scientific research on handgrip muscle fatigability performed by the Frailty in Ageing research department (see https://fria.research.vub.be/) and in collaboration with top-level international partners.

The eforto® system allows self-assessment of muscle fatigability and self-perceived fatigue in older adults and functions as a monitoring tool for intrinsic capacity. It is a small device, easy to use, and suitable for home measurements as well as hospital settings. When used correctly, the measurements cause no discomfort and can be performed repeatedly. The rubber bulb connects to a smartphone application that provides verbal test instructions to the participant. The app will guide the participant during the test and automatically provide motivational cues via audio. The test results are aggregated and stored in a cloud platform where the researcher can manage subjects, access the test data and export it for further analysis. The mobile app supports Dutch, French and English.

In a previous study, eforto® was clinically validated against a gold-standard pressure gauge in n=61 community-dwelling older adults, n=26 hospitalized geriatric patients and n=25 older hip fracture patients. Moreover, the usability and acceptance of eforto® self-monitoring (1 week) was demonstrated in a sample of n=30 community dwelling older persons aged between 83 and 95 years old. (paper submitted for publication in international peer-reviewed journal)

Procedures:

After the recruitment, a researcher will estimate whether the participant is eligible for the study during a eligibility check by a telephone call and legally capable to provide consent. After informed consent is given, baseline measurements will take place. These measurements will be reassessed after 6 months and 12 months. After an individual information session explaining how to use eforto®, the participant will be instructed to perform the eforto® measurements for 2 consecutive days per week for 12 months at home (if needed with assistance by an informal caregiver). Preferentially, the researcher will install the eforto® application on the smartphone of the participant. The home measurements will be continued for 12 months or until withdrawal of the participant. During the study, there will be a monthly telephone contact between participants and researchers in order to register technical problems, and self-reported changes in health situation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and over
* Living in the community (independently at home or at home assisted by an informal caregiver or in assistive housing)
* Being able to operate the basic functions of a smartphone (if needed with assistance by an informal caregiver): using a smartphone at least for calls and minimum 1 other application
* Understanding Dutch or French
* Simple Frail Scale score <3

Exclusion Criteria:

Being unable to participate in the assessments due to:

* Physical impairments (e.g. unable to stand up or walk)
* Cognitive impairments (unable to understand the test instructions and/or Mini Mental State Examination (MMSE) score <23/30)
* Functional disability of the dominant upper extremity (pare-sis/paralysis, tremor or recent surgery)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling older people aged 65 years and over.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Usability of the eforto® system | Week 1
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 2
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 3
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 4
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 5
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 6
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 7
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 8
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 9
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 10
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 11
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 12
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 13
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 14
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 15
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 16
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 17
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 18
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 19
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 20
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 21
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 22
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 23
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 24
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 25
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 26
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 27
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 28
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 29
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 30
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 31
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 32
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 33
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 34
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 35
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 36
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 37
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 38
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 39
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 40
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 41
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 42
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 43
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 44
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 45
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 46
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 47
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 48
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 49
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 50
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 51
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Usability of the eforto® system | Week 52
  A checklist of potential technical problems (11 questions) related to the eforto® system that can occur during the study. Options for answer: yes or no; if 'yes' => clarify the technical problem.
Feasibility of the eforto® system | End of the study (week 52)
  An self-reported questionnaire (12 questions) based on the technology acceptance model (the Unified Theory of Acceptance Use of Technology (UTAUT)). Options for answer: 1-5. 1 is 'Strongly disagree', 5 is 'Strongly agree'.

SECONDARY OUTCOMES:
The correlation between muscle fatigability and frailty status. | Baseline
  Muscle fatigability will be measured with the eforto® system (grip work, kPa*s). The frailty status will be assessed by the frailty assessments: a) Fried Criteria: consists of five components: unintentional weight loss, weakness, exhaustion (low energy level), slowness (slow gait) and low physical activity. This is operationalised through self-reported questions and non-invasive tests like grip strength using eforto® and timed 4-meter walking. Frailty is defined as having ≥3 of the 5 components, pre-frail participants have 1 or 2 components and robust participants have none of the components. b) Groningen Frailty Indicator: this is a 15-item self-reported questionnaire. Each positive answer is given a score of 1. A score of ≥4 indicates moderate to severe frailty.
The correlation between self-perceived fatigue and frailty status. | Baseline
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The Multidimensional Fatigue Inventory will be assessed in the context of self-perceived fatigue. The frailty status will be assessed by a) Fried Criteria: consists of 5 components: unintentional weight loss, weakness, exhaustion (low energy level), slowness (slow gait) and low physical activity. This is operationalised through self-reported questions and non-invasive tests. Frailty = having ≥3 of the 5 components, pre-frail = having 1 or 2 components and robust = having none of the components. b) Groningen Frailty Indicator: = 15-item self-reported questionnaire. Each positive answer is given a score of 1. A score of ≥4 indicates moderate to severe frailty.
The correlation between muscle fatigability and frailty status. | 6 months
  Muscle fatigability will be measured with the eforto® system (grip work, kPa*s). The frailty status will be assessed by the frailty assessments: a) Fried Criteria: consists of five components: unintentional weight loss, weakness, exhaustion (low energy level), slowness (slow gait) and low physical activity. This is operationalised through self-reported questions and non-invasive tests like grip strength using eforto® and timed 4-meter walking. Frailty is defined as having ≥3 of the 5 components, pre-frail participants have 1 or 2 components and robust participants have none of the components. b) Groningen Frailty Indicator: this is a 15-item self-reported questionnaire. Each positive answer is given a score of 1. A score of ≥4 indicates moderate to severe frailty.
The correlation between self-perceived fatigue and frailty status. | 6 months
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The Multidimensional Fatigue Inventory will be assessed in the context of self-perceived fatigue. The frailty status will be assessed by a) Fried Criteria: consists of 5 components: unintentional weight loss, weakness, exhaustion (low energy level), slowness (slow gait) and low physical activity. This is operationalised through self-reported questions and non-invasive tests. Frailty = having ≥3 of the 5 components, pre-frail = having 1 or 2 components and robust = having none of the components. b) Groningen Frailty Indicator: = 15-item self-reported questionnaire. Each positive answer is given a score of 1. A score of ≥4 indicates moderate to severe frailty.
The correlation between muscle fatigability and frailty status. | 12 months
  Muscle fatigability will be measured with the eforto® system (grip work, kPa*s). The frailty status will be assessed by the frailty assessments: a) Fried Criteria: consists of five components: unintentional weight loss, weakness, exhaustion (low energy level), slowness (slow gait) and low physical activity. This is operationalised through self-reported questions and non-invasive tests like grip strength using eforto® and timed 4-meter walking. Frailty is defined as having ≥3 of the 5 components, pre-frail participants have 1 or 2 components and robust participants have none of the components. b) Groningen Frailty Indicator: this is a 15-item self-reported questionnaire. Each positive answer is given a score of 1. A score of ≥4 indicates moderate to severe frailty.
The correlation between self-perceived fatigue and frailty status. | 12 months
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The Multidimensional Fatigue Inventory will be assessed in the context of self-perceived fatigue. The frailty status will be assessed by a) Fried Criteria: consists of 5 components: unintentional weight loss, weakness, exhaustion (low energy level), slowness (slow gait) and low physical activity. This is operationalised through self-reported questions and non-invasive tests. Frailty = having ≥3 of the 5 components, pre-frail = having 1 or 2 components and robust = having none of the components. b) Groningen Frailty Indicator: = 15-item self-reported questionnaire. Each positive answer is given a score of 1. A score of ≥4 indicates moderate to severe frailty.
The correlation between muscle fatigability and functional independency. | At baseline
  Muscle fatigability will be measured with the eforto® system (grip work, expressed in kPa*s). The functional independency will be assessed by the Katz Basic Activities of Daily Living (range of score: 6-24; a low score = high function, independent and a high score = low function, dependent) and the Lawton Instrumental Activities of Daily Living Scale (range of score: 9-27; a low score = low function, dependent and a high score = high function, independent).
The correlation between self-perceived fatigue and functional independency. | At baseline
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The participants will also complete the Multidimensional Fatigue Inventory in the context of self-perceived fatigue (also embedded in the eforto® system). The functional independency will be assessed by the Katz Basic Activities of Daily Living (range of score: 6-24; a low score = high function, independent and a high score = low function, dependent) and the Lawton Instrumental Activities of Daily Living Scale (range of score: 9-27; a low score = low function, dependent and a high score = high function, independent).
The correlation between muscle fatigability and functional independency. | 6 months
  Muscle fatigability will be measured with the eforto® system (grip work, expressed in kPa*s). The functional independency will be assessed by the Katz Basic Activities of Daily Living (range of score: 6-24; a low score = high function, independent and a high score = low function, dependent) and the Lawton Instrumental Activities of Daily Living Scale (range of score: 9-27; a low score = low function, dependent and a high score = high function, independent).
The correlation between self-perceived fatigue and functional independency. | 6 months
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The participants will also complete the Multidimensional Fatigue Inventory in the context of self-perceived fatigue (also embedded in the eforto® system). The functional independency will be assessed by the Katz Basic Activities of Daily Living (range of score: 6-24; a low score = high function, independent and a high score = low function, dependent) and the Lawton Instrumental Activities of Daily Living Scale (range of score: 9-27; a low score = low function, dependent and a high score = high function, independent).
The correlation between muscle fatigability and functional independency. | 12 months
  Muscle fatigability will be measured with the eforto® system (grip work, expressed in kPa*s). The functional independency will be assessed by the Katz Basic Activities of Daily Living (range of score: 6-24; a low score = high function, independent and a high score = low function, dependent) and the Lawton Instrumental Activities of Daily Living Scale (range of score: 9-27; a low score = low function, dependent and a high score = high function, independent).
The correlation between self-perceived fatigue and functional independency. | 12 months
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The participants will also complete the Multidimensional Fatigue Inventory in the context of self-perceived fatigue (also embedded in the eforto® system). The functional independency will be assessed by the Katz Basic Activities of Daily Living (range of score: 6-24; a low score = high function, independent and a high score = low function, dependent) and the Lawton Instrumental Activities of Daily Living Scale (range of score: 9-27; a low score = low function, dependent and a high score = high function, independent).
The correlation between muscle fatigability and quality of life. | At baseline
  Muscle fatigability will be measured with the eforto® system (grip work, kPa*s). The quality of life will be assessed by the self-reported questionnaires SarQol (short form), Eq-5D-5L, and Brief Resilience Scale.
The correlation between self-perceived fatigue and quality of life. | At baseline
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The participants will also complete the Multidimensional Fatigue Inventory in the context of self-perceived fatigue (also embedded in the eforto® system). The quality of life will be assessed by the self-reported questionnaires SarQol (short form), Eq-5D-5L, and Brief Resilience Scale.
The correlation between muscle fatigability and quality of life. | 6 months
  Muscle fatigability will be measured with the eforto® system (grip work, kPa*s). The quality of life will be assessed by the self-reported questionnaires SarQol (short form), Eq-5D-5L, and Brief Resilience Scale.
The correlation between self-perceived fatigue and quality of life. | 6 months
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The participants will also complete the Multidimensional Fatigue Inventory in the context of self-perceived fatigue (also embedded in the eforto® system). The quality of life will be assessed by the self-reported questionnaires SarQol (short form), Eq-5D-5L, and Brief Resilience Scale.
The correlation between muscle fatigability and quality of life. | 12 months
  Muscle fatigability will be measured with the eforto® system (grip work, kPa). The quality of life will be assessed by the self-reported questionnaires SarQol (short form), Eq-5D-5L, and Brief Resilience Scale.
The correlation between self-perceived fatigue and quality of life. | 12 months
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The participants will also complete the Multidimensional Fatigue Inventory in the context of self-perceived fatigue (also embedded in the eforto® system). The quality of life will be assessed by the self-reported questionnaires SarQol (short form), Eq-5D-5L, and Brief Resilience Scale.
The correlation between muscle fatigability and circulating inflammatory biomarkers. | At baseline
  Muscle fatigability will be measured with the eforto® system (grip work, kPa*s). The circulating inflammatory biomarkers will be measured by blood sampling:
  * 1x 3mL serum for determination of hsCRP.
  * Additional 1x 9mL EDTA and 1x 9mL serum tube will be obtained for determination of inflammation-related cyto/chemokines including IL1RA, IL6, IL10, TNFα, MCP1, suPAR and sRAGE.
The correlation between muscle fatigability and circulating inflammatory biomarkers. | 6 months
  Muscle fatigability will be measured with the eforto® system (grip work, kPa*s). The circulating inflammatory biomarkers will be measured by blood sampling:
  * 1x 3mL serum for determination of hsCRP.
  * Additional 1x 9mL EDTA and 1x 9mL serum tube will be obtained for determination of inflammation-related cyto/chemokines including IL1RA, IL6, IL10, TNFα, MCP1, suPAR and sRAGE.
The correlation between muscle fatigability and circulating inflammatory biomarkers. | 12 months
  Muscle fatigability will be measured with the eforto® system (grip work, kPa*s). The circulating inflammatory biomarkers will be measured by blood sampling:
  * 1x 3mL serum for determination of hsCRP.
  * Additional 1x 9mL EDTA and 1x 9mL serum tube will be obtained for determination of inflammation-related cyto/chemokines including IL1RA, IL6, IL10, TNFα, MCP1, suPAR and sRAGE.
The correlation between self-perceived fatigue and circulating inflammatory biomarkers. | At baseline
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The participants will also complete the Multidimensional Fatigue Inventory in the context of self-perceived fatigue (also embedded in the eforto® system). The circulating inflammatory biomarkers will be measured by blood sampling:
  * 1x 3mL serum for determination of hsCRP.
  * Additional 1x 9mL EDTA and 1x 9mL serum tube will be obtained for determination of inflammation-related cyto/chemokines including IL1RA, IL6, IL10, TNFα, MCP1, suPAR and sRAGE.
The correlation between self-perceived fatigue and circulating inflammatory biomarkers. | 6 months
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The participants will also complete the Multidimensional Fatigue Inventory in the context of self-perceived fatigue (also embedded in the eforto® system). The circulating inflammatory biomarkers will be measured by blood sampling:
  * 1x 3mL serum for determination of hsCRP.
  * Additional 1x 9mL EDTA and 1x 9mL serum tube will be obtained for determination of inflammation-related cyto/chemokines including IL1RA, IL6, IL10, TNFα, MCP1, suPAR and sRAGE.
The correlation between self-perceived fatigue and circulating inflammatory biomarkers. | 12 months
  Self-perceived fatigue will be measured with the eforto® system (2 self-perceived fatigue questions: Question 1: How fatigued are you feeling at this moment? Options for answer: 1-7. 1 is 'not tired', 7 is 'extremely tired'. Question 2: I fatigue quickly. Options for answer: 1-7. 1 is 'No, I don't agree', 7 is 'Yes, I agree'). The participants will also complete the Multidimensional Fatigue Inventory in the context of self-perceived fatigue (also embedded in the eforto® system). The circulating inflammatory biomarkers will be measured by blood sampling:
  * 1x 3mL serum for determination of hsCRP.
  * Additional 1x 9mL EDTA and 1x 9mL serum tube will be obtained for determination of inflammation-related cyto/chemokines including IL1RA, IL6, IL10, TNFα, MCP1, suPAR and sRAGE.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rasmussen LJH, Caspi A, Ambler A, Danese A, Elliott M, Eugen-Olsen J, Hariri AR, Harrington H, Houts R, Poulton R, Ramrakha S, Sugden K, Williams B, Moffitt TE. Association Between Elevated suPAR, a New Biomarker of Inflammation, and Accelerated Aging. J Gerontol A Biol Sci Med Sci. 2021 Jan 18;76(2):318-327. doi: 10.1093/gerona/glaa178. PMID 32766674
- [Background] Frimat M, Teissier T, Boulanger E. Is RAGE the receptor for inflammaging? Aging (Albany NY). 2019 Sep 8;11(17):6620-6621. doi: 10.18632/aging.102256. Epub 2019 Sep 8. No abstract available. PMID 31494645
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Bautmans I, Mets T. A fatigue resistance test for elderly persons based on grip strength: reliability and comparison with healthy young subjects. Aging Clin Exp Res. 2005 Jun;17(3):217-22. doi: 10.1007/BF03324600. PMID 16110735
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Beaudart C, Biver E, Reginster JY, Rizzoli R, Rolland Y, Bautmans I, Petermans J, Gillain S, Buckinx F, Dardenne N, Bruyere O. Validation of the SarQoL(R), a specific health-related quality of life questionnaire for Sarcopenia. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):238-244. doi: 10.1002/jcsm.12149. Epub 2016 Oct 22. PMID 27897430
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] van Hooff ML, Geurts SA, Kompier MA, Taris TW. "How fatigued do you currently feel?" Convergent and discriminant validity of a single-item fatigue measure. J Occup Health. 2007 May;49(3):224-34. doi: 10.1539/joh.49.224. PMID 17575403
- [Background] Alberts M, Smets EM, Vercoulen JH, Garssen B, Bleijenberg G. ['Abbreviated fatigue questionnaire': a practical tool in the classification of fatigue]. Ned Tijdschr Geneeskd. 1997 Aug 2;141(31):1526-30. Dutch. PMID 9543741
- See also: FORTO-aal site — https://forto-aal.eu/
- See also: Frailty in ageing research group VUB site — https://fria.research.vub.be/